CLINICAL TRIAL: NCT00414687
Title: An Explorative, Open-Label, Multicenter, Randomized, Parallel-Group Comparative Study of Safety, Tolerability, and the Clinical Effects of Iloprost Inhalation in Patients With Primary or Secondary Pulmonary Hypertension Over 2 Years
Brief Title: Aerosolized Randomized Iloprost Study II (AIR - II) Long-Term Safety, Tolerability, and Clinical Effects of Iloprost Inhalation in Patients With Primary or Secondary Pulmonary Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Schering Pharma AG
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 90427; 300341
Record Dates: First submitted 2006-12-20; First posted 2006-12-21 (Estimated); Last update posted 2009-05-15 (Estimated); Status verified 2009-05

CONDITIONS: Hypertension, Pulmonary
Keywords: Primary or secondary Pulmonary hypertension; Iloprost; Inhaled; Long-term treatment
MeSH Terms: conditions — Hypertension, Pulmonary; Respiratory Aspiration | interventions — Iloprost

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Ventavis (Iloprost, BAYQ6256)

INTERVENTIONS:
Drug: Ventavis (Iloprost, BAYQ6256)

SUMMARY:
The purpose of this study is to determine whether the study drug is effective in the long-term treatment of primary or secondary pulmonary hypertension

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.

Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients
* Secondary pulmonary hypertension
* Mean pulmonary artery pressure equal or above 40 mmHg or primary pulmonary hypertension with a pressure equal or above 30 mmHg while resting during appropriate conventional treatment
* Written informed consent after having been duly informed about all diagnostic and therapeutic measures involved in the study

Exclusion Criteria:

* Clinical Instability at baseline
* Pulmonary venous obstruction
* Global respiratory insufficiency
* Obstructive ventilation disorders, Interstitial pulmonary disease
* Cerebrovascular events
* Myocardial infarction or major cardiac surgery within 3 months prior to baseline
* Bleeding disorders or bleeding risk
* Severe hepatic insufficiency or renal insufficiency
* Malignant diseases
* HIV positive
* Pregnancy, female patients of child-bearing potential without adequate contraception and nursing mothers
* Congenital or acquired valvular defects and myocardial function disorders not related to pulmonary hypertension
* Prior pulmonary embolism
* Collagenosis
* Pulmonary arterial or valvular stenosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 1998-07; Study Completion 2001-05 (Actual)

PRIMARY OUTCOMES:
Tolerability: Adverse events (AE) and safety variables, Variables to describe clinical effects: NYHA class, Walking distance (6-min walk), Mahler Dyspnea Index, EuroQoL, Karnofsky Index, Hemodynamic and gas exchange
Mortality and lung/heart-lung transplantation, Acute effects of iloprost inhalation on hemodynamics and gas exchange

SECONDARY OUTCOMES:
Overall clinical tolerability of the long-term use of iloprost aerosol
Serious Adverse Events and deaths
Effect of long-term administration of inhaled iloprost on mortality and transplantation
Exercise capacity
Acute effect of inhaled iloprost on hemodynamics and gas exchange
Effects of long-term administration of inhaled iloprost on hemodynamics and gas exchange
Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer

REFERENCES:
- [Derived] Olschewski H, Hoeper MM, Behr J, Ewert R, Meyer A, Borst MM, Winkler J, Pfeifer M, Wilkens H, Ghofrani HA, Nikkho S, Seeger W. Long-term therapy with inhaled iloprost in patients with pulmonary hypertension. Respir Med. 2010 May;104(5):731-40. doi: 10.1016/j.rmed.2010.01.008. Epub 2010 Feb 11. PMID 20153158